CLINICAL TRIAL: NCT01982448
Title: A Randomized Phase II Study of Preoperative Cisplatin Versus Paclitaxel in Patients With Triple Negative Breast Cancer: Evaluating the Homologous Recombination Deficiency (HRD) Biomarker
Brief Title: Cisplatin vs Paclitaxel for Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Myriad Genetics, Inc. (Industry); Translational Breast Cancer Research Consortium (Other)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principal Invesitigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-383; TBCRC030 (Other: Translational Breast Cancer Research Consortium)
Record Dates: First submitted 2013-10-28; First posted 2013-11-13 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: TRIPLE NEGATIVE BREAST CANCER; CISPLATIN; PACLITAXEL
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Cisplatin (Experimental): Cisplatin given by IV infusion at a dose of 75 mg/m2 every 3 weeks (1 cycle) for 4 cycles as preoperative chemotherapy. Participants with inadequate clinical response after 12 weeks (as judged either clinically or radiologically by a provider) were able to crossover to an alternative provider-selected preoperative chemotherapy regimen. Definitive breast surgery following no later than 42 days after administration of last chemotherapy.
  Interventions: Drug: Cisplatin
- Arm B: Paclitaxel (Experimental): Paclitaxel given by IV infusion at a dose of 80 mg/m2 weekly for 12 weeks (4 cycles) as neoadjuvant chemotherapy. Participants with inadequate clinical response after 12 weeks (as judged either clinically or radiologically by a provider) were able to 'crossover' to an alternative provider-selected preoperative chemotherapy regimen. Definitive breast surgery following no later than 42 days after administration of last chemotherapy.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Cisplatin
  Other Names: Platinol ®-AQ
  Arms: Arm A: Cisplatin
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Arm B: Paclitaxel

SUMMARY:
This is a phase II study randomizing patients with stage I with T1 > 1.5 cm, stage II or III triple negative breast cancer (TNBC) to preoperative cisplatin versus paclitaxel. The study is designed to evaluate the ability of the Homologous Recombination Deficiency (HRD) assay to predict pathologic response to preoperative chemotherapy.

DETAILED DESCRIPTION:
Cisplatin and paclitaxel are active in triple-negative breast cancer (TNBC). Despite different mechanisms of action, effective predictive biomarkers to preferentially inform drug selection have not been identified. The homologous recombination deficiency (HRD) assay (Myriad Genetics, Inc.) detects impaired double-strand DNA break repair and may identify patients with BRCA1/2-proficient tumors that are sensitive to DNA-targeting therapy. The primary objective of TBCRC 030 was to detect an association of HRD with pathologic response (residual cancer burden (RCB)-0/1) to singleagent cisplatin or paclitaxel. This prospective phase II study enrolled patients with germline BRCA1/2 wild-type/unknown stage I-III TNBC in a 12-week randomized study of preoperative cisplatin or paclitaxel. The HRD assay was carried out on baseline tissue; positive HRD was defined as a score >=33. Crossover to an alternative chemotherapy was offered if there was inadequate response.

ELIGIBILITY:
Inclusion Criteria: 1. Participants must meet the following criteria on screening examination to be eligible to participate in the study 2. Pathologic documentation of invasive breast cancer by biopsy (FNA alone is not adequate). 3. AJCC clinical stage I with T1 > 1.5 cm, stage II or III invasive breast cancer. 4. Participants with multicentric or bilateral disease are eligible if at least one lesion meets stage eligibility criteria for the study and no tumor is HER2-positive. 5. Tumors must be HER2 negative defined as HER2 0 or 1+ by immunohistochemistry (IHC) assays and /or lack of gene amplification by FISH defined as a ratio < 2 on invasive tumor by local review. 6. ER and PgR status by IHC must be known. Tumor must be ER and PR negative (≤5% staining) by local review. 7. Known BRCA1/2 (BReast CAncer) status is not required for study entry. However patients known to have a germline deleterious BRCA1/2 mutation should be encouraged to consider a preoperative trial specifically designed for BRCA1/2 carriers, if available. 8. Breast imaging should include imaging of the ipsilateral axilla. For subjects with a clinically positive axilla, a needle aspiration, core biopsy or SLN procedure will be performed to confirm the presence of metastatic disease in the lymph nodes. For patients with a clinically negative axilla, baseline assessment of the axilla will be performed at the discretion of the treating investigator. For patients with pathologically positive axillary lymph nodes prior to preoperative therapy, a level I and II lymph node dissection at the time of definitive surgery is recommended. 9. Patients with a prior history of contra-lateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer within the last 5 years. 10. Women ≥ 18 years of age. 11. ECOG performance status ≤1 (see Appendix A). 12. Laboratory Evaluation 1) Absolute neutrophil count (ANC) ≥ 1,500 / mm3 2) Platelet count ≥ 100,000/ mm3 3) Bilirubin ≤ 1.5x upper limit of normal (ULN), for patients with Gilbert syndrome, direct bilirubin will be measured instead of total bilirubin 4) ALT, AST ≤3.0 x ULN ALK Phos <2.5 x ULN 5) Creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 cc/min 6) Hemoglobin ≥ 9 mg/dl 7) Use of an effective means of contraception is required in subjects of childbearing potential since study agents are known to be teratogenic. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. 8) Ability to understand and the willingness to sign a written informed consent document 9) Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy and did not receive prior chemotherapy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. 10) Patient must be willing to undergo mandatory research biopsy and blood draw. Prior to biopsy procedures patients must be able to be off medications that could increase the risk of bleeding Exclusion Criteria: 1. Participants with axillary adenopathy only are not eligible for this study. 2. Prior chemotherapy: Prior non-taxane or platinum containing chemotherapy will be allowed if the prior exposure was at least 5 years ago and the exposure is thought not to potentially interact with the primary outcome of the trial or put the patient at undue risk, and should be reviewed with study PI on a case by case basis. 3. Any prior treatment for the current breast cancer, including chemotherapy, hormonal therapy, radiation or experimental therapy. 4. Ipsilateral breast recurrence, unless prior treatment consisted of excision alone for DCIS or breast conserving treatment and hormonal therapy for DCIS or invasive breast cancer. 5. Ongoing use of any other investigational or study agents. 6. Peripheral neuropathy of any etiology > grade 1 (NCI CTCAE Version 4.0- Appendix B) 7. Significant hearing loss that would prevent cisplatin administration. 8. Renal dysfunction for which exposure to cisplatin would be unsafe or require cisplatin dose modification (i.e., Cre > 1.5 mg/dl or GFR < 60 cc/min).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-04; Primary Completion 2019-01 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (20):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Indiana University- Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - Memorial Sloan Kettering Cancer Center-Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center-Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center-Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center-West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center-Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center-Sleepy Hollow, Sleepy Hollow, New York
  - University of North Carolina- Lineberger Cancer Center, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Universtiy of Pittsburgh- Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Cancer Alliance at EvergreenHealth, Kirkland, Washington
  - University of Washignton, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mayer EL, Abramson V, Jankowitz R, Falkson C, Marcom PK, Traina T, Carey L, Rimawi M, Specht J, Miller K, Stearns V, Tung N, Perou C, Richardson AL, Componeschi K, Trippa L, Tan-Wasielewski Z, Timms K, Krop I, Wolff AC, Winer EP. TBCRC 030: a phase II study of preoperative cisplatin versus paclitaxel in triple-negative breast cancer: evaluating the homologous recombination deficiency (HRD) biomarker. Ann Oncol. 2020 Nov;31(11):1518-1525. doi: 10.1016/j.annonc.2020.08.2064. Epub 2020 Aug 13. PMID 32798689
- [Derived] Nader-Marta G, Chu X, Mukhopadhyay S, Abramson VG, Brufsky A, Stringer-Reasor EM, Dent SF, Traina TA, Carey LA, Rimawi MF, Specht JM, Miller KD, Santa-Maria CA, Dasgupta T, Kurt BB, DeMeo M, Krop IE, Tung NM, Schnitt SJ, Tayob N, Mayer EL. Prognostic value of visually and computationally assessed tumor-infiltrating lymphocytes in early-stage triple-negative breast cancer (TBCRC-030). J Natl Cancer Inst. 2026 Jan 1;118(1):141-149. doi: 10.1093/jnci/djaf289. PMID 41075163
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32798689/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2014 through January 2018
Period: Preoperative Chemotherapy
Arm/Group | Arm A: Cisplatin | Arm B: Paclitaxel
Started | 75 | 72
Eligible & Treated | 72 | 70
Evaluable for Safety (Participants who completed at least one cycle of neoadjuvant chemotherapy were evaluable for adverse events.) | 72 | 68
Completed | 72 | 67
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Ineligible Prior to Starting Therapy | 1 | 0
Not completed — Hypersensitivity during cycle 1 so therapy stopped | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: Definitive Breast Surgery
Arm/Group | Arm A: Cisplatin | Arm B: Paclitaxel
Started | 72 | 67
Evaluable for Response by Homologous Recombination Deficiency (HRD) (Participants with baseline diagnostic tissue for HRD analysis.) | 56 | 48
Completed | 72 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Cisplatin | Arm B: Paclitaxel | Total
Number analyzed (Participants) | 75 | 72 | 147
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 82] | 53.5 [30 to 73] | 53 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 72 | 147
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 4 | 11
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 60 | 51 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 72 | 147
BRCA1/2 Status [Count of Participants; unit: Participants]
  Germline/somatic intact | 69 | 71 | 140
  Germline and/or somatic mutation | 6 | 1 | 7
Clinical lymph node status [Count of Participants; unit: Participants]
  Positive | 29 | 26 | 55
  Negative | 46 | 46 | 92
Homologous Recombination Deficiency (HRD) Status [Count of Participants; unit: Participants] — HRD status was determined with baseline diagnostic tissue using the HRD assay (Myriad Genetics, Inc.; required minimum 100 mm2 of tumor tissue) which detects impaired double-strand DNA break repair. The positive threshold for HRD was a score >/= 33. Population: The analysis population is comprised of all participants with evaluable tissue for HRD analysis and who completed definitive breast surgery.
  Participants
    number analyzed (Participants) | 56 | 48 | 104
    HRD High (+) Status | 39 | 35 | 74
    HRD Low (-) Status | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Response by HR-deficiency (HRD) Status
Description: Pathologic response was assessed using the MD Anderson residual cancer burden (RCB) method (Symmans et al. JCO 2007). Responders are defined as RCB 0/1 and non-responders as RCB 2/3. Participants who crossed over due inadequate clinical response after 12 weeks were counted as non-responders. HRD status was determined with baseline diagnostic tissue using the HRD assay (Myriad Genetics, Inc.; required minimum 100 mm2 of tumor tissue) which detects impaired double-strand DNA break repair. The positive threshold for HRD was a score >/= 33.
Time Frame: Evaluated after definitive breast surgery, up to 4-5 months from enrollment.
Population: The analysis population is comprised of all participants with evaluable tissue for HRD analysis and who completed definitive breast surgery.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Cisplatin With HRD+: Cisplatin given by IV infusion at a dose of 75 mg/m2 every 3 weeks (1 cycle) for 4 cycles as preoperative chemotherapy. Participants with inadequate clinical response after 12 weeks (as judged either clinically or radiologically by a provider) were able to crossover to an alternative provider-selected preoperative chemotherapy regimen. Definitive breast surgery following no later than 42 days after administration of last chemotherapy. HRD+ (score >/=33)
- Arm A: Cisplatin With HRD-: Cisplatin given by IV infusion at a dose of 75 mg/m2 every 3 weeks (1 cycle) for 4 cycles as preoperative chemotherapy. Participants with inadequate clinical response after 12 weeks (as judged either clinically or radiologically by a provider) were able to crossover to an alternative provider-selected preoperative chemotherapy regimen. Definitive breast surgery following no later than 42 days after administration of last chemotherapy. HRD- (score <33)
- Arm B: Paclitaxel With HRD+: Paclitaxel given by IV infusion at a dose of 80 mg/m2 weekly for 12 weeks (4 cycles) as neoadjuvant chemotherapy. Participants with inadequate clinical response after 12 weeks (as judged either clinically or radiologically by a provider) were able to crossover to an alternative provider-selected preoperative chemotherapy regimen. Definitive breast surgery following no later than 42 days after administration of last chemotherapy. HRD+ (score >/=33)
- Arm B: Paclitaxel With HRD-: Paclitaxel given by IV infusion at a dose of 80 mg/m2 weekly for 12 weeks (4 cycles) as neoadjuvant chemotherapy. Participants with inadequate clinical response after 12 weeks (as judged either clinically or radiologically by a provider) were able to crossover to an alternative provider-selected preoperative chemotherapy regimen. Definitive breast surgery following no later than 42 days after administration of last chemotherapy. HRD- (score <33)
Arm/Group | Arm A: Cisplatin With HRD+ | Arm A: Cisplatin With HRD- | Arm B: Paclitaxel With HRD+ | Arm B: Paclitaxel With HRD-
Number analyzed (Participants) | 39 | 17 | 35 | 13
Participants
  Responder (RCB-0/1) | 9 | 2 | 10 | 4
  Non-Responder (RCB-2/3 or crossover) | 30 | 15 | 25 | 9
Statistical Analysis 1: Comparison: Arm A: Cisplatin With HRD+ vs Arm A: Cisplatin With HRD-; In the Cisplatin treated patients, the relationship between HRD status and pathologic response was conducted by arm using a univariate logistic regression model and a likelihood ratio test with a one-sided type I error of alpha 0.05. Assuming 12.5% unevaluable, prevalence of HR deficiency 60%, 70 evaluable patients per in a given arm, there is ~80% power to detect a response rate of 52% in HR-deficient patients vs a 16% in HR non-deficient patients, corresponding to the Odds Ratio 5.7; Test type: Superiority; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.39 to 23.68] — Association between HRD status and pathologic response was measured by the odds ratio (OR)
Statistical Analysis 2: Comparison: Arm B: Paclitaxel With HRD+ vs Arm B: Paclitaxel With HRD-; In the Paclitaxel treated patients, the relationship between HRD status and pathologic response was conducted by arm using a univariate logistic regression model and a likelihood ratio test with a one-sided type I error of alpha 0.05. Assuming 12.5% unevaluable, prevalence of HR deficiency 60%, 70 evaluable patients per in a given arm, there is ~80% power to detect a response rate of 37% in HR-deficient patients vs a 16% in HR non-deficient patients, corresponding to the Odds Ratio 0.62; Test type: Superiority; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.19 to 4.95]

2. Secondary Outcome: Number With Pathologic Complete Response (pCR) by HR-deficiency (HRD) Status
Description: Pathologic response was assessed using the MD Anderson residual cancer burden (RCB) method (Symmans et al. JCO 2007). pCR is defined as RCB-0. HRD status was determined with baseline diagnostic tissue using the HRD assay (Myriad Genetics, Inc.; required minimum 100 mm2 of tumor tissue) which detects impaired double-strand DNA break repair. The positive threshold for HRD was a score >/= 33.
Time Frame: Evaluated after definitive breast surgery, up to 4-5 months from enrollment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Cisplatin With HRD+ | Arm A: Cisplatin With HRD- | Arm B: Paclitaxel With HRD+ | Arm B: Paclitaxel With HRD-
Number analyzed (Participants) | 39 | 17 | 35 | 13
Participants
  pCR | 5 | 1 | 5 | 3
  No pCR | 34 | 16 | 30 | 10
Statistical Analysis 1: Comparison: Arm A: Cisplatin With HRD+ vs Arm A: Cisplatin With HRD-; Test type: Superiority; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.23 to 118.07]
Statistical Analysis 2: Comparison: Arm B: Paclitaxel With HRD+ vs Arm B: Paclitaxel With HRD-; Test type: Superiority; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.09 to 4.14]

3. Secondary Outcome: Number of Pathologic Response
Description: as for outcome 1
Time Frame: Evaluated after definitive breast surgery, up to 4-5 months from enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Cisplatin | Arm B: Paclitaxel
Number analyzed (Participants) | 72 | 67
Participants
  Responder (RCB-0/1) | 19 | 15
  Non-responder (RCB-2/3 or crossover) | 53 | 52

4. Secondary Outcome: Number With Pathologic Response
Description: as for outcome 1
Time Frame: Evaluated after definitive breast surgery, up to 4-5 months from enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Cisplatin | Arm B: Paclitaxel
Number analyzed (Participants) | 72 | 67
Participants
  pCR | 11 | 8
  Non-pCR | 61 | 59

5. Secondary Outcome: Positive Predictive Value (PPV) of HRD Score
Description: Pathologic response was assessed using the MD Anderson residual cancer burden (RCB) method (Symmans et al. JCO 2007). Responders are defined as RCB 0/1 and non-responders as RCB 2/3. Participants who crossed over due inadequate clinical response after 12 weeks were counted as non-responders. HRD status was determined with baseline diagnostic tissue using the HRD assay (Myriad Genetics, Inc.; required minimum 100 mm2 of tumor tissue) which detects impaired double-strand DNA break repair. The positive threshold for HRD was a score >/= 33. PPV was calculated as the probability of pathological response among the HRD positive group.
Time Frame: Evaluated after definitive breast surgery, up to 4-5 months from enrollment.
Measure: Number; unit: probability
Arm/Group | Arm A: Cisplatin | Arm B: Paclitaxel
Number analyzed (Participants) | 39 | 35
probability | .231 | .286

ADVERSE EVENTS:
Time Frame: AE data collected every cycle from the time of the first dose of study treatment, through the study 12 weeks of treatment until 30 days after removal from study or death, whichever occurs first. Therefore, AEs were observed up to 4 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Groups:
- Paclitaxel: Paclitaxel will be given as an IV infusion at a dose of 80mg/m2 weekly x 12 weeks (4 cycles).
- Cisplatin: Cisplatin will be given by IV at 75 mg/m2 every 3 weeks, 4 cycles.
Arm/Group | Paclitaxel | Cisplatin
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/67
Serious Adverse Events (participants affected / at risk) | 11/72 | 19/67
Other Adverse Events (participants affected / at risk) | 72/72 | 67/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel (N=72) | Cisplatin (N=67)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 8
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Nasal congestion (Metabolism and nutrition disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel (N=72) | Cisplatin (N=67)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 21
Tinnitus (Ear and labyrinth disorders) | 1 | 5
Vertigo (Ear and labyrinth disorders) | 0 | 2
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 37 | 33
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 2
Mitral valve disease (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 3 | 2
Chills (General disorders) | 1 | 2
Edema limbs (General disorders) | 4 | 3
Fatigue (General disorders) | 51 | 55
Fever (General disorders) | 1 | 3
Flu like symptoms (General disorders) | 2 | 2
Infusion related reaction (General disorders) | 8 | 0
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 9 | 3
Pain (General disorders) | 10 | 5
General disorders and administration site conditions - Other (General disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 6 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 14 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 3 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 11 | 3
Hypothyroidism (Endocrine disorders) | 1 | 6
Endocrine disorders - Other (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Bloating (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 19 | 31
Diarrhea (Gastrointestinal disorders) | 23 | 16
Dry mouth (Gastrointestinal disorders) | 5 | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 10 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10 | 12
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 31 | 57
Oral dysesthesia (Gastrointestinal disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 13
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 | 4
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 1
Bladder infection (Infections and infestations) | 0 | 1
Breast infection (Infections and infestations) | 1 | 1
Bronchial infection (Infections and infestations) | 1 | 0
Gum infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 1
Upper respiratory infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Vaginal infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 3 | 2
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 16 | 6
Alkaline phosphatase increased (Investigations) | 3 | 10
Aspartate aminotransferase increased (Investigations) | 14 | 8
Blood bilirubin increased (Investigations) | 2 | 1
Cardiac troponin T increased (Investigations) | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 1
Cholesterol high (Investigations) | 9 | 3
Creatinine increased (Investigations) | 1 | 10
Hemoglobin increased (Investigations) | 1 | 2
Lymphocyte count decreased (Investigations) | 6 | 0
Lymphocyte count increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 24 | 39
Platelet count decreased (Investigations) | 3 | 16
Weight gain (Investigations) | 2 | 1
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 25 | 29
Investigations - Other (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 23
Hyponatremia (Metabolism and nutrition disorders) | 6 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 7
Obesity (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 2
Metabolism and nutrition disorders - Other, (Metabolism and nutrition disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Growth suppression (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 | 6
Akathisia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 9
Dysgeusia (Nervous system disorders) | 15 | 11
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 25 | 18
Hypersomnia (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 7 | 1
Peripheral motor neuropathy (Nervous system disorders) | 11 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 40 | 10
Presyncope (Nervous system disorders) | 0 | 2
Nervous system disorders - Other (Nervous system disorders) | 2 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Nervous system disorders) | 1 | 0
Blurred vision (Eye disorders) | 3 | 1
Conjunctivitis (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 2 | 2
Flashing lights (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 2 | 0
Watering eyes (Eye disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 24 | 17
Depression (Psychiatric disorders) | 14 | 7
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 24 | 15
Libido decreased (Psychiatric disorders) | 0 | 1
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute kidney injury (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Bladder spasm (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Surgical and medical procedures - Other (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 12 | 10
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0
Menopause (Reproductive system and breast disorders) | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2 | 2
Flushing (Vascular disorders) | 2 | 2
Hot flashes (Vascular disorders) | 13 | 8
Hypertension (Vascular disorders) | 22 | 19
Hypotension (Vascular disorders) | 1 | 1
Lymphedema (Vascular disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 0 | 2
Vascular disorders - Other (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT01982448/Prot_SAP_000.pdf